CLINICAL TRIAL: NCT03348579
Title: Hospital Acquired and Ventilator Associated Pneumonia : Impact of the New French Guidelines on Patients Care and Outcomes.
Brief Title: Hospital-acquired Pneumonia in Intensive Care Unit
Acronym: PNEUMOCARE
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0434
Record Dates: First submitted 2017-11-16; First posted 2017-11-21 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2017-11

CONDITIONS: Hospital Acquired Pneumonia; Ventilator-Associated Pneumonia; Sepsis; Pneumonia
Keywords: Intensive care unit; Pneumonia; Ventilator associated; Hospital acquired pneumonia; Guidelines
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated; Sepsis; Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The before period: The before period (control phase) will consist of all consecutive patients admitted to the participating ICUs before the national guidelines publication concerning hospital-acquired pneumonia.
  Interventions: Other: Guidelines publication and application
- The second period: Intensive care units are randomized in two groups:
  Standard training: The centers will receive the text of the recommendation electronically. The principal investigator of each center will then train doctors, interns, nurses and physiotherapists to the use of these recommendations (team leader). A computer presentation common to all the centers will be used and a communication strategy vis-à-vis the other caregivers of the investigative services will be put in place. All doctors, interns and nurses must have attended this theoretical training during the awareness phase.
  Interventions: Other: Guidelines publication and application; Other: Targeted experience feedback
- The third and final period: The third and final period will consist of all consecutive patients admitted to the participating ICUs after the formal training.
  Interventions: Other: Guidelines publication and application

INTERVENTIONS:
Other: Guidelines publication and application — Passing recommendations on using the guidelines in the intensive care units
Other: Targeted experience feedback — Targeted experience feedback": On top of the standard training, the centers receive an analysis of the evolution of the practices of their center and the future of their patients between phases 1 and 2, as well as these same values for the data set. The centers are then called to conduct a meeting to determine their priority improvement points based on this audi
  Groups: The second period

SUMMARY:
hospital-acquired pneumonia are a common disease in intensive care unit. The prevention, the diagnosis and the treatment of hospital acquired pneumonia are a frequent challenge. Nevertheless it seems that there are great differences in standard of care between hospitals. The investigators hypothesized that medical education and implementation of evidence-base guidelines can reduce the duration of mechanical ventilation in patients presenting of hospital acquired pneumonia

DETAILED DESCRIPTION:
The before period (phase 1) will consist of all consecutive patients admitted to the participating ICUs before the national guidelines publication concerning healthcare associated pneumonia.

The second period (phase 2) will consist of all consecutive patients admitted to the participating ICUs after the publication of the national guidelines publication concerning healthcare associated pneumonia.

Afterward, an interphase will occur during which all physicians, residents, physiotherapists and nurses will receive a formal training for the processes and procedures related to the new guidelines published in september 2017.

In the intervention group, on top of the standard training, the centers receive an analysis of the evolution of the practices of their center and the future of their patients between phases 1 and 2, as well as these same values for the data set. The centers are then called to conduct a meeting to determine their priority improvement points based on this audit.

The third and final period (phase 3) will consist of all consecutive patients admitted to the participating ICUs after the formal training.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years ; IGS-II score > 15 ; Hospital stay >= 3 days

Exclusion Criteria:

* Community-acquired pneumonia, pregnant women, refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients hospitalized in intensive care units with a hospital stay greater than 72 hours and a GIs-II greater than or equal to 15.
Sampling Method: Non-Probability Sample
Enrollment: 1850 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Unit length of stay | 28 days
  Duration of ICU hospitalization Safety Issue: NA

SECONDARY OUTCOMES:
Intensive Care Unit free-days at day 28 | 28 days
  The number of days from day 1 to day 28 on which a patient is alive outside of intensive care unit Safety Issue
Hospital-acquired pneumonia | 28 days
  definition based on the appearance of a new infiltrate or changes in an existing infiltrate on chest X-ray associated with any two of the following clinical signs: body temperature >38°C, leucocytosis >12,000/ml or leukopenia <4000/ml, and purulent pulmonary secretions that were associated with a positive quantitative or semi-quantitative bacteriological culture of a respiratory tract sample.
Composite measure of compliance to guidelines | 28 days
  defined as the total number of performed eligible measures divided by the total number of measures for which each patient was eligible
Empirical treatment failure | 28 days
  Defined as one or more pathogen involved in the pneumonia is not susceptible to the antibiotics used empirically

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Roquilly, PH, Principal Investigator — Nantes University Hospital; Marc Leone, Principal Investigator — AP-HM
Locations (1):
- CHU de NANTES, Nantes, France

REFERENCES:
- [Derived] Roquilly A, Chanques G, Lasocki S, Foucrier A, Fermier B, De Courson H, Carrie C, Danguy des Deserts M, Gakuba C, Constantin JM, Lagarde K, Holleville M, Blidi S, Sossou A, Cailliez P, Monard C, Oudotte A, Mathieu C, Bourenne J, Isetta C, Perrigault PF, Lakhal K, Rouhani A, Asehnoune K, Guerci P, Tran Dinh A, Chousterman B, Cupaciu A, Dahyot-Fizelier C, Bellier R, Au Duong J, Mansour A, Morel J, Beauplet G, Vibet MA, Feuillet F, Sebille V, Leone M. Implementation of French Recommendations for the Prevention and the Treatment of Hospital-acquired Pneumonia: A Cluster-randomized Trial. Clin Infect Dis. 2021 Oct 5;73(7):e1601-e1610. doi: 10.1093/cid/ciaa1441. PMID 32970811